CLINICAL TRIAL: NCT02527135
Title: Evaluating Feasibility and Potential Impact of Text Messages on HIV Awareness Among Young Women in Rural Kenya: a Pilot Study
Brief Title: Text Messaging to Improve HIV Testing Among Young Women in Kenya
Acronym: T2T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Grand Challenges Canada (Other); National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Njambi Njuguna, Dr, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 49533-EJ; D43TW009580 (NIH); S4 0254-01 (Other Grant/Funding Number: Grand Challenges Canada)
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: HIV Infection
Keywords: SMS; Text messages; Young women; HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioural (Experimental): Intervention arm receiving weekly HIV sensitization text messages
  Interventions: Behavioral: Weekly HIV sensitization text messages
- Control (No Intervention): No weekly messages were sent to this group

INTERVENTIONS:
Behavioral: Weekly HIV sensitization text messages — Weekly HIV sensitization text messages with option to text back up to 3 times per week for additional messages. Message topics included pregnancy, condoms, sexually transmitted infections, contraceptives, anal sex and personal risk of HIV. All messages ended with the phrase "Get tested for HIV".
  Arms: Behavioural

SUMMARY:
The purpose of this study is to determine whether regularly scheduled HIV sensitization text messages (SMS) are effective in increasing HIV testing rates among young women in Kenya.

DETAILED DESCRIPTION:
In Kenya, women have higher rates of infection (6.9%) than men (4.4%) and young women aged 15-24 years are over three times more likely to be infected than young men of the same age group. HIV testing and counseling remains critical to identifying new infections and preventing the spread of HIV but many young women do not test and still continue to engage in high risk behavior.

HIV programs have begun to leverage mobile phones and text messages to increase the reach and scale of interventions. Kenya currently has 32.2 million mobile phone subscribers, representing a 79.2% country penetration. Text messages have been used successfully in Kenya for marketing purposes and have even been demonstrated to increase antiretroviral (ART) adherence. Despite advances in mobile-based applications to improve issues in health, none of these health applications have yet been able to reach the scale of mobile phone-based financial products in Kenya.

Given the potential synergies of text message use and need for HIV testing, a randomized quasi-experimental study was conducted to test whether weekly text messages encouraging HIV testing and improving HIV awareness would increase HIV testing, enhance HIV risk perception and reduce high risk behaviour among young women 18-24 years old in a predominantly rural region in Kenya.

Women in the intervention arm received access to a suite of HIV sensitization text messages sent weekly to increase their awareness of HIV and encourage them to test with the option of texting back for more information to a maximum of three times per week. Women in the control arm did not receive these messages. All women were followed up for six months with monthly SMS surveys collecting data on their HIV testing practices, sexual behaviour and risk perception.

ELIGIBILITY:
Inclusion Criteria:

* Own a mobile phone which they don't share and which operates on a telecom provider supported by our SMS platform
* Be HIV uninfected (by self report) or not know their HIV status
* Report not having tested for HIV in the preceding 12 months
* Know how to send and receive SMS
* Must consent to the study
* Have regular access to electricity for charging a cell phone

Exclusion Criteria:

* Did not consent to the study
* Did not meet inclusion criteria

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
First HIV test | End of study (6 months after enrollment)
  Time to first reported HIV test will be compared between the two study arms

SECONDARY OUTCOMES:
Reported sexual behaviour patterns | End of study (6 months after enrollment)
  Sexual behaviour data (number of new sexual partners, concurrent sexual partnerships and number of sex acts where condoms are used) was collected via a text message survey monthly during study follow up and responses will be compared between the two study arms
Self perception of risk | End of study (6 months after enrollment)
  Self perception of HIV risk in both arms will be compared against HIV testing habits and sexual partnerships

CONTACTS AND LOCATIONS:
Overall Officials: Njambi Njuguna, MBChB,MPH, Principal Investigator — University of Washington; Kenyatta National Hospital
Locations (1):
- Partners in Health and Research Development (PHRD), Nairobi, Nairobi County, Kenya